CLINICAL TRIAL: NCT03922763
Title: Does a Fixed Inclination Humeral Cut in Anatomic Total Shoulder Arthroplasty Effectively Recreate Normal Anatomy: A Prospective Randomized Trial
Brief Title: Fixed Inclination Humeral Cut
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019Laz
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Shoulder Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anatomically-matched cut (Active Comparator)
  Interventions: Procedure: Anatomical cut
- Cutting guide (Active Comparator)
  Interventions: Procedure: Cutting guide

INTERVENTIONS:
Procedure: Anatomical cut — Surgeon-derived cut based on patient's anatomy
  Arms: Anatomically-matched cut
Procedure: Cutting guide — Angle cut at 132.5 degrees based on cutting guide
  Arms: Cutting guide

SUMMARY:
The purpose of the present study is to determine if a standard humeral cut using a fixed neck shaft angled prosthesis for patients undergoing anatomic TSA is able to restore normal glenohumeral relationships as compared to a variable neck shaft angle prosthesis.

ELIGIBILITY:
Inclusion Criteria:

1. patients 18 years or older
2. primary glenohumeral osteoarthritis
3. intact rotator cuff
4. primary anatomic shoulder arthroplasty

Exclusion Criteria:

1. revision arthroplasty
2. reverse shoulder arthroplasty candidates
3. cognitive or behavioral problems which would preclude informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-02 (Actual); Primary Completion 2020-02-02 (Estimated); Study Completion 2020-05-02 (Estimated)

PRIMARY OUTCOMES:
Radriographic measurements | x-rays taken day of surgery
  x-rays will be measured by 3 independent surgeons to measure restoration to natural anatomy following total shoulder replacement

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States